CLINICAL TRIAL: NCT00002345
Title: Phase IV Study on the Safety and Efficacy of Megace Oral Suspension in HIV-Positive Females
Brief Title: The Safety and Effectiveness of Megace in HIV-Infected Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 025C; MEG169-93.007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Anorexia; Cachexia; HIV Infections
Keywords: Megestrol; Acquired Immunodeficiency Syndrome; Anorexia; Cachexia; Suspensions
MeSH Terms: conditions — Anorexia; Cachexia; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Megestrol Acetate

INTERVENTIONS:
Drug: Megestrol acetate

SUMMARY:
To further evaluate the safety of megestrol acetate (Megace) oral suspension in the treatment of anorexia and cachexia in HIV-positive women. To compare the effectiveness of 2 doses of Megace by measurement of weight gain, appetite grade, and other parameters at 12 and 24 weeks.

DETAILED DESCRIPTION:
Patients are randomized to receive 1 of 2 doses of Megace oral suspension daily for 24 weeks; at 12 weeks, those receiving the lower dose who have not gained 5 pounds over baseline or had appetite improvement to good or excellent are escalated to the higher dose. Patients are evaluated at 4-week intervals. Dose may be adjusted to maintain a desired weight.

ELIGIBILITY:
Inclusion Criteria

Patient must have:

* HIV infection.
* Evidence of HIV wasting syndrome that includes anorexia (appetite fair or poor) and weight loss >= 10 percent of pre-illness body weight.
* Perception of weight loss as a detriment.
* Life expectancy of at least 24 weeks.

Prior Medication:

Allowed:

* Megestrol acetate for weight gain at a dose < 400 mg for < 60 days, provided therapy was discontinued at least 3 months prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Poorly controlled hypertension.
* Heart failure.
* Deep vein thrombosis.
* Uncontrolled severe diarrhea.
* Treatable active current infection (excluding chronic low-grade opportunistic infections).
* Unable to intake food.
* Impaired digestive/absorptive function.

Concurrent Medication:

Excluded:

* Initiation during the study of any therapy to treat HIV or anorexia/cachexia (other than study drug).

Patients with the following prior conditions are excluded:

* Hospitalization for or exacerbation of illness associated with weight loss within the past 2 weeks.
* Participation in other investigational drug studies within the past month.
* Previous abnormal mammogram (if 35-40 years of age) or abnormal mammogram within the past year (if over 40 years of age).

Prior Medication:

Excluded:

* New antiviral therapy within the past 8 weeks.
* Medications to promote weight gain (e.g., corticosteroid, dronabinol) within the past 2 months.
* Megestrol acetate within the past 3 months. IV drug abuse not treated for at least 4 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Univ of California - Davis Med Ctr / CARES, Sacramento, California
  - Yale Univ Med School, New Haven, Connecticut
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Miriam Hosp, Providence, Rhode Island